CLINICAL TRIAL: NCT03687099
Title: Immunological and Functional Characterization of Cellular Population CD45+ Infiltrating Human Glioblastoma
Acronym: GLIOBLASTOMES
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2018_843_0011
Record Dates: First submitted 2018-05-17; First posted 2018-09-27 (Actual); Last update posted 2020-07-16 (Actual); Status verified 2020-07

CONDITIONS: Glioblastoma
Keywords: Glioblastoma; CD45; Lymphocytes; Microglia; Macrophage
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — Histological samples from 10 GBM removed from patients with long-term survival and 10 GBM removed from patients with short-term survival

SUMMARY:
Despite advances in neurosurgery , radiotherapy and chemotherapy, the median survival in GBM patients is only 15 months from diagnosis. Immunotherapy by checkpoint inhibitors (PD1 /PDL-1) appears as a promising treatment for many cancers. However, first clinical results are disappointing for GBM. An hypothesis is the immunosuppressive activity from infiltrating non-tumor cells. Conversion of non-tumor cells from an immunosuppressive to an immuno-activating phenotype could be attempted in a therapeutic perspective.

DETAILED DESCRIPTION:
An important and constant infiltration of cells marked with CD45 has been observed in 77 GBM studied for the prognostic value of PDL1 and IL17 infiltration (in association with Pr Ghiringhelli ; INSERM ; Dijon) . However, CD45 is present at the surface of all leucocytes. The purpose of this project is to better characterize the nature and functionality of the CD45+ cells that infiltrate GBM (lymphocytes and their sub-types, macrophages, microglial cells). Formalin-fixed paraffin-embedded GBM samples will be studied. A panel of immune cell antibody will be used for the immuno-histological (IH) study. Furthermore, the investigator will compare these data with those obtained by the nanoString technology, a multiplexed measurement of gene expression.

ELIGIBILITY:
Inclusion Criteria:

* Formalin-fixed paraffin-embedded GBM samples from tumor bank of the pathological laboratory of the University Hospital of Amiens-Picardie.
* Histologic diagnosis of a glioblastoma according to the WHO classification of central nervous system
* Radical surgical removal in order to have enough histological material and to homogenize the main prognostic factor that is the surgical removal.
* Patients with more than 18 years old.
* Patients informed who have signed a consent form for using the tumor for research purposes without personal benefit. If patients were died, absence of objection known for the anonymous use of the tumor for scientific purpose.
* Be insured under one social security system.
* Committee for the protection of persons approval.

Exclusion Criteria:

* Relapsed GBM
* Other brain tumors.
* Medical, psychological or social conditions not allowing the comprehension of the conduct of the study for patients able to give their opinion.
* Patient under curatorship.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Histological samples of GBM
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2018-04-30 (Actual); Primary Completion 2019-11-08 (Actual); Study Completion 2019-11-08 (Actual)

PRIMARY OUTCOMES:
number of cells which express CD45 in the immunological environment from GBM. | 1
  number of cells which express CD45 in the immunological environment from GBM, with using NanoString/RNAseq (NGS) and immunohistology

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens-Picardie, Amiens, France